CLINICAL TRIAL: NCT01881919
Title: A Double-Blind, Cross-Over, Placebo-Controlled Study Evaluating the Effect of Quercetin 500 mg Tablets on Blood Uric Acid in Healthy Males
Brief Title: Effect of Quercetin Supplements on Healthy Males: a Four-Week Randomized Cross-Over Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Yuanlu Shi, PhD Candidate, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEEC12-019
Record Dates: First submitted 2013-06-07; First posted 2013-06-20 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Hyperuricemia; Gout; Kidney Calculi; Diabetes; Cardiovascular Disease
Keywords: Functional Food
MeSH Terms: conditions — Hyperuricemia; Gout; Kidney Calculi; Diabetes Mellitus; Cardiovascular Diseases | interventions — Therapeutics; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Treatment (Experimental): Daily intake of Quercetin supplement 500mg tablet for 28 days with meal (breakfast preferred.)
  Interventions: Dietary Supplement: Treatment
- Placebo (Placebo Comparator): Daily intake of Placebo (lactose) tablet for 28 days with meal (breakfast preferred)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Treatment — Address: Nature's Best, Century Place, Tunbridge Wells, Kent, TN2 3BE Phone:+44(0)1892 552030 Email:info@naturesbest.co.uk
  Other Names: Quercetin dihydrate 500 mg tablet; Brand: Nature's Best; Batch Number:114501; Serial Number: 5055148404901
  Arms: Treatment
Dietary Supplement: Control — Address: Fagron GmbH&Co. KG, 22885 Barsbuttel, Germany Phone: +49(0)4067067680
  Other Names: Placebo: lactose tablet; Brand: Fagron; Serial Number: PZN-0921071; Batch Number:1208D001A
  Arms: Placebo

SUMMARY:
The purpose of this study was to test the effect of chronic consumption of Quercetin 500 mg tablets on blood uric acid and other biomarkers in adult males.

DETAILED DESCRIPTION:
The main goal of the research is to determine the long term effects of daily supplementation of quercetin, a compound naturally and normally present in food, on the chemical composition (uric acid ii and glucose) of blood and urine and on blood pressure, of healthy males.

Six of the volunteers will collect urine after consuming a standard meal made from fresh onion and after quercetin supplement intake, in the same way, with 3 days washout before each. The urine collected here will be analysed to check that the supplement is equivalent to the food. Stage 2 will only be conducted with supplement and placebo.

Healthy male volunteers with higher (than average) blood uric acid will be selected and will be asked to consume a standard supplement/placebo added to their own diet for 4 weeks per phase. Two arms are separated by 4 weeks resting period: quercetin supplement and placebo. Blood and urine samples will be taken every other week to detect any changes of uric acid and other biomarkers.

----- i) Quercetin is found in a variety of foods including apples, berries, brassica vegetables, capers, grapes, onions, shallots, tea, and tomatoes, as well as many seeds, nuts, flowers, barks, and leaves.

ii) Uric acid, a compound found in both in the human body and urine, is produced by the breakdown of purines, which are nitrogen-containing compounds in substances such as nucleic acids (DNA). They enter the circulation from digestion of certain foods, drinks (alcoholic beverages like beer and wine) or from normal breakdown and turnover of cells in the body. Most uric acid is removed by the kidneys and disposed of in the urine; the remainder is excreted in the stool.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Plasma Uric Acid > 300 micro Mole/L
* Generally Healthy

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 30 kg/m² or <18.5 kg/m²
* Unable or unwilling to comply with the protocol, or likely to leave the study before its completion.
* Who would undertake important change in physical exercise or vigorous sport competitions during the study period.
* regularly drink more than 3 units of alcohol every day
* smokers
* have history of treated hyperuricemia, gout and/ or kidney stone
* have intestinal disorders

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Risk of getting hyperuricemia assessed by the measure of plasma uric acid. | Fasting blood samples are taken on day 1, day 15 and day 29 of each arm
  The change of plasma uric acid level from day 1 on day 15 and day 29 of each arm.

SECONDARY OUTCOMES:
Kidney excretion of uric acid: urinary uric acid level | 24 h urine samples are collected on day 14 and 28 of each arm and volume is recorded
  Difference in 24-h urinary uric acid level at 14 days and 28 days between arms
Blood pressure | Blood pressure is measured on day 1 and 29 of each arm
  To monitor the compliance of subject.
Blood glucose | Fasted blood samples are collected on day 1, 15, 29 of each arm
  The change of plasma glucose level from the baseline at day 15 and day 29 of each arm.
Metabolomic and metabonomic profiling of blood plasma | Fasting blood samples are taken on day 1, day 15 and day 29 of each arm
  1H NMR (proton nuclear magnetic resonance )

OTHER OUTCOMES:
Urinary excretion of quercetin | 24 h urine will be collected on day 14 and 28 of each arm and volume is recorded
  To monitor the compliance of subject.
Subject Body Weight | weight is measured on day 1 and 29 of each arm
  To monitor the compliance of subject.
Subject Height | Height is measured on day 1 and 29 of each arm
  To monitor the compliance of subject.
Life style maintenance | Recall Questionnaires about the past 28 days are required on day 1 and 29 of each arm.
  To monitor the compliance of subject.
Primary health assessment | Recall Questionnaires about history of certain disease, routine medication / supplements, allergies and exercise/diet practice at enrollment
  To set baseline for maintaining lifestyle and routine medicine for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williamson, PhD, Study Chair — University of Leeds; Yuanlu Shi, PhD Candidate, Principal Investigator — University ofLeeds
Locations (1):
- School of Food Science and Nutrition, Leeds, West Yorkshire, United Kingdom